CLINICAL TRIAL: NCT01084317
Title: Evaluation of the Delay in Asthma Diagnosis in Children From the Lodz Region After the Program for Prevention of Allergic Diseases
Brief Title: Evaluation of the Delay in Asthma Diagnosis in Children From the Lodz Region
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Professor, Medical University of Lodz
Other Study IDs: RNN/603/09/KB
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Bronchial Asthma
Keywords: asthma; children; delay in asthma diagnosis
MeSH Terms: conditions — Asthma | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- asthmatic children: patients under 18 age, with newly diagnosed asthma
  Interventions: Other: medical documentation and telephone interview

INTERVENTIONS:
Other: medical documentation and telephone interview — medical documentation analysis supplemented by telephone interview conducted with parents of the child

SUMMARY:
The aim of the research is to assess the duration of a delay in asthma diagnosis in children after the Program for Prevention of Allergic Diseases. Risk factors for delayed diagnosis of asthma in children will also be assessed. This study will answer the question of whether this ratio depends on the time, which indirectly proves that it can be changed by local intervention programs. Prove lasting effects of the Program may contribute to planning further local interventions focused on improving medical care for patients with bronchial asthma in the Lodz region, and reduce social costs associated with this disease.

DETAILED DESCRIPTION:
The object of this study is asthma, the most common chronic childhood disease. The disease has become epidemic in developed countries and also in Poland. The percentage of children suffering from bronchial asthma in Lodz is one of the highest in the country (8.5%. Bronchial asthma in children of Lodz is a real challenge not only for doctors but also for public health professionals. This study is to assess the long-term effects of innovation on a national scale Prevention Program of Allergic Diseases, which was carried out in 2000-2003 in the region of Lodz. This Program has given many positive effects, most of all, improvement in the diagnosis of allergic diseases, availability of medical specialists and reduction the number of hospitalizations because of the disease exacerbation.

The aim of the research is to assess the duration of a delay in asthma diagnosis in children after the Program for Prevention of Allergic Diseases. Risk factors for delayed diagnosis of asthma in children will also be assessed. This study will answer the question of whether this ratio depends on the time, which indirectly proves that it can be changed by local intervention programs. Prove lasting effects of the Program may contribute to planning further local interventions focused on improving medical care for patients with bronchial asthma in the Lodz region, and reduce social costs associated with this disease.

Subject of study are patients under 18 age, with newly diagnosed asthma, who were under care in Allergy Clinic in Copernicus Hospital in Lodz in 2004-2009. Selected clinic is the largest pediatric allergy center in the region and was also the largest center participating in the Program for Prevention of Allergic Diseases and the only center, which analyzed the delay in asthma diagnosis among patients. Children's medical documentation will be analyzed as far as following data were concerned: demographic data, anthropometric parameters, information about family history of atopic diseases, asthma symptoms (cough, dyspnoea, wheezing, reducing physical activity, and recurrent respiratory infections) and symptoms of other atopic diseases in both the current and in the past. In addition, information will be collected on the child's family situation, housing conditions and the presence of animals in the house. Data obtained from the children's medical documentation will be supplemented by telephone interview conducted with parents of the child. The group of patients with underdiagnosed asthma will be classified as children who experienced frequent wheezing (at least 4 episodes per year) and 1 major criterium (positive family history of allergic diseases or symptoms of atopic as infants) or two smaller criteria (symptoms of food allergies, the increased number of eosinophilic cells in the peripheral blood or wheezing without infection). For each child the time from appearance of asthma symptoms (according to the API - asthma predictive index) to diagnose the disease by a specialist will be set. This time will be defined as duration of undiagnosed asthma. Due to the fact that the delay in asthma diagnosis is dependent on the patient's age, the analysis will be carried out in four groups separated on the basis of the upper and lower quartiles of respondents age.

ELIGIBILITY:
Inclusion Criteria:

* patients under 18 age, with newly diagnosed asthma

Exclusion Criteria:

* patients under 18 age, without newly diagnosed asthma

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients under 18 age, with newly diagnosed asthma,
Sampling Method: Probability Sample
Enrollment: 907 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
duration of a delay in asthma diagnosis in children | 5 years
  The duration of a delay in asthma diagnosis in children after the Program for Prevention of Allergic Diseases

CONTACTS AND LOCATIONS:
Overall Officials: Włodzimierz Stelmach, MD, PhD, Study Chair — Department of Social and Preventive Medicine, Medical University of Lodz, Poland; Iwona Stelmach, MD,PhD,Prof., Study Director — Department of Pediatrics and Allergy, N. Copernicus Hospital, Medical University of Lodz, Poland; Ewa Bąk, Master of Sc, Principal Investigator — Department of Social and Preventive Medicine, Medical University of Lodz, Poland
Locations (1):
- Department of Social and Preventive Medicine, Medical University of Lodz, Poland, Department of Pediatrics and Allergy, N. Copernicus Hospital, Medical University of Lodz, Poland, Lodz, Poland